CLINICAL TRIAL: NCT03384745
Title: A Phase 2b Randomized, Double-blind, Placebo Controlled, Multi-center 12-week Study With an Additional 40-week Follow-up Assessment of Efficacy, Safety and Tolerability of M1095 in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis
Brief Title: A Phase 2b Study of the Efficacy, Safety, and Tolerability of M1095 (Sonelokimab) in Subjects With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bond Avillion 2 Development LP (Industry)
Collaborators: Avillion LLP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AV002
Record Dates: First submitted 2017-12-20; First posted 2017-12-27 (Actual); Results first posted 2021-08-02 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — sonelokimab; secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- M1095 (Sonelokimab) 30mg (Experimental): M1095, 30 mg, given at Week 0, 2, 4, 8, 12 and every four weeks.
  Interventions: Drug: M1095 (Sonelokimab)
- M1095 (Sonelokimab) 60mg (Experimental): M1095, 60 mg, given at Week 0, 2, 4, 8, 12 and every four weeks.
  Interventions: Drug: M1095 (Sonelokimab)
- M1095 (Sonelokimab) 120mg - regimen 1 (Experimental): M1095, 120 mg, given at Week 0, 2, 4, 8, 12 and every eight weeks.
  Interventions: Drug: M1095 (Sonelokimab)
- M1095 (Sonelokimab) 120mg - regimen 2 (Experimental): M1095, 120 mg, given at Week 0, 2, 4, 6, 8, 10, 12 and every four weeks.
  Interventions: Drug: M1095 (Sonelokimab)
- Placebo / M1095 (Sonelokimab) 120mg (Placebo Comparator): Placebo, given at Week 0, 1, 2, 3, 4, 6, 8 and 10, then M1095, 120mg, given at Week 12, 14, 16, and every four weeks.
  Interventions: Drug: M1095 (Sonelokimab); Drug: Placebo
- Secukinumab (Active Comparator): Secukinumab, 300mg, given at Week 0, 1, 2, 3, 4, 8, 12 and every four weeks.
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: M1095 (Sonelokimab) — M1095 (Sonelokimab) is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
  Other Names: Sonelokimab
  Arms: M1095 (Sonelokimab) 120mg - regimen 1; M1095 (Sonelokimab) 120mg - regimen 2; M1095 (Sonelokimab) 30mg; M1095 (Sonelokimab) 60mg; Placebo / M1095 (Sonelokimab) 120mg
Drug: Placebo — Placebo contains no active drug.
  Arms: Placebo / M1095 (Sonelokimab) 120mg
Drug: Secukinumab — Secukinumab is a human immunoglobulin G1 (IgG1) monoclonal antibody that selectively binds IL-17A.
  Other Names: Cosentyx®
  Arms: Secukinumab

SUMMARY:
This is a multi-center phase 2b study in subjects with moderate to severe chronic plaque-type psoriasis. Approximately 300 subjects will be enrolled at approximately 60 investigator sites in North America and Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 18 and 75 years of age.
2. Moderate to severe plaque-type psoriasis for at least 6 months.
3. Subject is a candidate for systemic biologic therapy.
4. Subject has IGA ≥3, involved body surface area (BSA) ≥10%, and PASI ≥12 at screening and at baseline.
5. Subject is able to comply with the study procedures.
6. Subject must provide informed consent.

Exclusion Criteria (Main):

1. Non-plaque type psoriasis, drug-induced psoriasis, or other skin conditions (e.g., eczema). (Psoriatic arthritis is allowed).
2. Other medical conditions, including planned surgery or active infection / history of infection, as defined in the study protocol. Subjects will be screened for tuberculosis and hepatitis B / hepatitis C.
3. Laboratory abnormalities at screening, as defined in the study protocol.
4. Prior use of systemic or topical treatments for psoriasis, as defined in the study protocol.
5. Prior use of any compound targeting IL-17, more than two biologic therapies, ustekinumab within 6 months, or TNF targeting therapies within 12 weeks.
6. History of suicidal thoughts within 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Kim Papp, Principal Investigator — Probity Medical Research Inc
Locations (55):
- United States (11):
  - Investigative Site, Birmingham, Alabama
  - Investigative Site, San Diego, California
  - Investigative Site, DeLand, Florida
  - Investigative Site, Sandy Springs, Georgia
  - Investigative Site, St Louis, Missouri
  - Investigative Site, Albuquerque, New Mexico
  - Investigative Site, New York, New York
  - Investigative Site, Bexley, Ohio
  - Investigative Site, Dallas, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, San Antonio, Texas
- Bulgaria (3):
  - Investigative Site, Dupnitsa
  - Investigative Site, Sofia
  - Investigative Site, Varna
- Canada (10):
  - Investigative Site, Edmonton, Alberta
  - Investigative Site, Surrey, British Columbia
  - Investigative Site, Markham, Ontario
  - Investigative Site, North Bay, Ontario
  - Investigative Site, Oakville, Ontario
  - Investigative Site, Ottawa, Ontario
  - Investigative Site, Richmond Hill, Ontario
  - Investigative Site, Waterloo, Ontario
  - Investigative Site, Windsor, Ontario
  - Investigative Site, Québec, Quebec
- Czechia (7):
  - Investigative Site, Brno
  - Investigative Site, Náchod
  - Investigative Site, Nový Jičín
  - Investigative Site, Ostrava
  - Investigative Site, Pardubice
  - Investigative Site, Prague
  - Investigative Site, Uherské Hradiště
- Germany (13):
  - Investigative Site, Augsburg
  - Investigative Site, Berlin
  - Investigative Site, Bochum
  - Investigative Site, Darmstadt
  - Investigative Site, Frankfurt am Main
  - Investigative Site, Friedrichshafen
  - Investigative Site, Hamburg
  - Investigative Site, Kiel
  - Investigative Site, Mahlow
  - Investigative Site, Mainz
  - Investigative Site, Osnabrück
  - Investigative Site, Quedlinburg
  - Investigative Site, Schwerin
- Hungary (5):
  - Investigative Site, Budapest
  - Investigative Site, Kecskemét
  - Investigative Site, Orosháza
  - Investigative Site, Szeged
  - Investigative Site, Szolnok
- Poland (6):
  - Investigative Site, Katowice
  - Investigative Site, Lublin
  - Investigative Site, Poznan
  - Investigative Site, Siedlce
  - Investigative Site, Skierniewice
  - Investigative Site, Warsaw

REFERENCES:
- [Result] Papp KA, Weinberg MA, Morris A, Reich K. IL17A/F nanobody sonelokimab in patients with plaque psoriasis: a multicentre, randomised, placebo-controlled, phase 2b study. Lancet. 2021 Apr 24;397(10284):1564-1575. doi: 10.1016/S0140-6736(21)00440-2. PMID 33894834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were adults aged 18-75 years with stable, moderate to severe plaque type psoriasis for >6 months prior to randomisation, and who were candidates for systemic biologic therapy.
Groups:
- M1095 30mg: M1095, 30 mg, given at Week 0, 2, 4, 8, 12 and every four weeks.
  Subjects with IGA>1 at Week 12 were escalated to receive M1095, 120mg
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- M1095 60mg: M1095, 60 mg, given at Week 0, 2, 4, 8, 12 and every four weeks.
  Subjects with IGA>1 at Week 12 were escalated to receive M1095, 120mg
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- M1095 120mg - Regimen 1: M1095, 120 mg, given at Week 0, 2, 4, 8, 12 and every eight weeks.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- M1095 120mg - Regimen 2: M1095, 120 mg, given at Week 0, 2, 4, 6, 8, 10, 12 and every four weeks.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- Placebo / M1095 120mg: Placebo, given at Week 0, 1, 2, 3, 4, 6, 8 and 10, then M1095, 120mg, given at Week 12, 14, 16, and every four weeks.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
  Placebo: Placebo contains no active drug.
Period: Placebo Controlled Induction (W0 - W12)
Arm/Group | M1095 30mg | M1095 60mg | M1095 120mg - Regimen 1 | M1095 120mg - Regimen 2 | Placebo / M1095 120mg | Secukinumab
Started | 52 | 52 | 53 | 51 | 52 | 53
Completed | 52 | 51 | 50 | 49 | 49 | 51
Not Completed | 0 | 1 | 3 | 2 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Period: Maintenance/Escalation (W12-W24)
Arm/Group | M1095 30mg | M1095 60mg | M1095 120mg - Regimen 1 | M1095 120mg - Regimen 2 | Placebo / M1095 120mg | Secukinumab
Started | 52 | 51 | 50 | 49 | 49 | 51
Completed | 52 | 51 | 49 | 47 | 47 | 51
Not Completed | 0 | 0 | 1 | 2 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1 | 0 | 0
Period: Response Assess/Dose Hold (W24-W48)
Arm/Group | M1095 30mg | M1095 60mg | M1095 120mg - Regimen 1 | M1095 120mg - Regimen 2 | Placebo / M1095 120mg | Secukinumab
Started | 52 | 51 | 49 | 47 | 47 | 51
Completed | 51 | 48 | 45 | 43 | 46 | 49
Not Completed | 1 | 3 | 4 | 4 | 1 | 2
Not completed — Adverse Event | 1 | 1 | 3 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- M1095 30mg: M1095, 30 mg, given at Week 0, 2, 4, 8, 12 and every four weeks.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- M1095 60mg: M1095, 60 mg, given at Week 0, 2, 4, 8, 12 and every four weeks.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- Total: Total of all reporting groups
Arm/Group | M1095 30mg | M1095 60mg | M1095 120mg - Regimen 1 | M1095 120mg - Regimen 2 | Placebo / M1095 120mg | Secukinumab | Total
Number analyzed (Participants) | 52 | 52 | 53 | 51 | 52 | 53 | 313
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (13.4) | 46.9 (12.3) | 44.1 (13.1) | 43.2 (13.2) | 45.9 (12.9) | 47.5 (13.8) | 46.0 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 43 | 34 | 39 | 38 | 228
  Male | 16 | 14 | 10 | 17 | 13 | 15 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 3 | 2 | 1 | 2 | 15
  Not Hispanic or Latino | 48 | 49 | 50 | 49 | 51 | 51 | 298
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 2 | 1 | 8 | 2 | 6 | 3 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 2 | 2 | 1 | 6
  White | 49 | 48 | 45 | 47 | 44 | 49 | 282
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 7 | 9 | 11 | 9 | 12 | 11 | 59
  Hungary | 6 | 8 | 6 | 4 | 5 | 4 | 33
  United States | 10 | 7 | 6 | 5 | 3 | 5 | 36
  Czechia | 13 | 14 | 13 | 8 | 16 | 16 | 80
  Poland | 8 | 8 | 7 | 13 | 5 | 10 | 51
  Bulgaria | 7 | 4 | 8 | 10 | 9 | 5 | 43
  Germany | 1 | 2 | 2 | 2 | 2 | 2 | 11
Height (cm) [Mean (Standard Deviation); unit: centimetres] — Population: Height was not captured for one subject at baseline.
  centimetres
    number analyzed (Participants) | 52 | 52 | 53 | 50 | 52 | 53 | 312
    (all) | 173 (10.4) | 173 (9.60) | 174 (9.89) | 173 (11.2) | 173 (10.1) | 172 (9.98) | 173 (10.2)
Weight at baseline (kg) [Mean (Standard Deviation); unit: kilograms] | 92.0 (19.0) | 91.5 (20.6) | 89.0 (18.3) | 93.0 (22.6) | 91.3 (24.1) | 90.3 (22.4) | 91.2 (21.1)
Prior biological use (actual) [Count of Participants; unit: Participants] — Prior biological use included treatment with ustekinumab (stopping at least six months prior to randomization), tumour necrosis factor (TNF) targeting therapies (stopping at least 12 weeks prior to randomization), or investigational therapies (stopping at least 12 weeks, or 5 half lives, whichever is the longer, prior to randomization).
  Subjects treated with more than 2 biological therapies as above were excluded from the study.
  Subjects receiving prior treatment at any time with any compound (marketed or investigational) targeting interleukin-17 were excluded from the study.
  Participants
    Yes | 9 | 10 | 9 | 7 | 8 | 7 | 50
    No | 43 | 42 | 44 | 44 | 44 | 46 | 263
Duration of psoriasis (years) [Mean (Standard Deviation); unit: years] | 20.0 (13.6) | 19.7 (12.8) | 15.8 (12.9) | 18.0 (11.7) | 16.3 (12.1) | 20.2 (13.6) | 18.3 (12.8)
Presence of psoriatic arthritis [Count of Participants; unit: Participants]
  Yes | 2 | 5 | 7 | 6 | 3 | 2 | 25
  No | 50 | 47 | 46 | 45 | 49 | 51 | 288
Investigator's Global Assessment (IGA) at baseline [Count of Participants; unit: Participants] — Investigator's Global Assessment is a rating scale for overall psoriatic disease. Assessment ranges from 0 (clear of psoriasis), 1 (almost clear), 2 (mild), 3 (moderate) or 4 (severe).
  Participants
    3 | 38 | 37 | 39 | 40 | 41 | 38 | 233
    4 | 14 | 15 | 14 | 11 | 11 | 15 | 80
Psoriasis Area and Severity Index (PASI) at baseline [Mean (Standard Deviation); unit: units on a scale] — The Psoriasis Area and Severity Index (PASI) combines assessments of the extent of body-surface area involvement in four anatomical regions (head, trunk, arms, legs) and the severity of desquamation, erythema and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72.0 for the most severe disease.
  units on a scale | 20.3 (7.91) | 20.7 (9.34) | 21.1 (8.38) | 20.6 (7.15) | 20.5 (6.89) | 21.7 (8.80) | 20.8 (8.08)
Percentage of total Body Surface Area (BSA) affected at baseline [Mean (Standard Deviation); unit: % of body surface area affected] — The percentage of total Body Surface Area (BSA) affected by plaque-type psoriasis was estimated from the percentages of areas affected, including head, trunk, upper limbs and lower limbs.
  % of body surface area affected | 26.0 (15.7) | 24.8 (15.6) | 25.3 (14.8) | 26.4 (12.8) | 26.2 (16.7) | 28.1 (16.1) | 26.1 (15.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Investigator's Global Assessment (IGA) Score of 0 or 1
Description: The primary endpoint is achievement of an IGA score of 0 or 1 at Week 12, with an IGA reduction of at least 2 points from baseline. The percentage of subjects in the Intent to Treat (ITT) Analysis Set with an IGA score of 0 or 1 at Week 12 will be used to compare treatment arms. IGA is the Investigator's Global Assessment of the extent of psoriasis, with 0 = clear of psoriasis, 1 = almost clear, 2 = mild psoriasis, 3 = moderate psoriasis, and 4 = severe psoriasis (the worst assessment on this scale). Higher scores in the IGA indicate a worse outcome.
Time Frame: Week 12, as compared to Week 0 (baseline)
Measure: Count of Participants; unit: Participants
Groups:
- M1095 30mg: M1095, 30 mg, given at Week 0, 2, 4, and 8 weeks.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- M1095 60mg: M1095, 60 mg, given at Week 0, 2, 4, and 8 weeks.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- M1095 120mg - Normal Load Group: M1095, 120 mg, given at Week 0, 2, 4, and 8 weeks.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- M1095 120mg - Augmented Load Group: M1095, 120 mg, given at Week 0, 2, 4, 6, 8, and 10 weeks.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- Placebo: Placebo, given at Week 0, 1, 2, 3, 4, 6, 8 and 10 weeks.
  Placebo: Placebo contains no active drug.
- Secukinumab: Secukinumab, 300mg, given at Week 0, 1, 2, 3, 4, and 8 weeks.
  Secukinumab: Secukinumab is a human immunoglobulin G1 (IgG1) monoclonal antibody that selectively binds IL-17A.
Arm/Group | M1095 30mg | M1095 60mg | M1095 120mg - Normal Load Group | M1095 120mg - Augmented Load Group | Placebo | Secukinumab
Number analyzed (Participants) | 52 | 52 | 53 | 51 | 52 | 53
Participants | 25 | 44 | 41 | 45 | 0 | 41
Statistical Analysis 1: Comparison: M1095 30mg vs Placebo; Null hypotheses were tested at Week 12 (individual M1095 treatment arms would not be different from placebo with respect to achievement of IGA scores of 0 or 1). The primary analysis was based on the intent-to-treat (ITT) population using a non-responder imputation (NRI) for missing values. Primary treatment comparisons versus placebo were made with the two-sided Cochran-Mantel-Haenszel (CMH) test stratified by actual prior biologic use (yes/no) and body weight (<=90; >90kg); Test type: Superiority — A sample size of 300 subjects has 99% power to detect a statistically significant difference between any treatment arm and placebo in the IGA score of 0 or 1 rate at Week 12, with a two-sided, unadjusted type I error of 0.05. Calculations assume IGA score 0 or 1 rates >88% for study drug and <=7% for placebo; p < 0.0001, Cochran-Mantel-Haenszel; At Week 12, none (0.0% [95% CI 0.0-6.8]) of the 52 participants in the placebo group had an IGA score of 0 or 1 versus 25 (48.1% [34.0-62.4], p<0.0001) of 52 participants in the M1095 30mg treatment group. Odds ratio could not be calculated due to the placebo group containing no responders
Statistical Analysis 2: Comparison: M1095 60mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; At Week 12, none (0.0% [95% CI 0.0-6.8]) of the 52 participants in the placebo group had an IGA score of 0 or 1 versus 44 (84.6% [71.9-93.1], p<0.0001) of 52 participants in the M1095 60mg treatment group. Odds ratio could not be calculated due to the placebo group containing no responders
Statistical Analysis 3: Comparison: M1095 120mg - Normal Load Group vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; At Week 12, none (0.0% [95% CI 0.0-6.8]) of the 52 participants in the placebo group had an IGA score of 0 or 1 versus 41 (77.4% [63.8-87.7], p<0.0001) of 53 participants in the M1095 120mg normal load treatment group. Odds ratio could not be calculated due to the placebo group containing no responders
Statistical Analysis 4: Comparison: M1095 120mg - Augmented Load Group vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; At Week 12, none (0.0% [95% CI 0.0-6.8]) of the 52 participants in the placebo group had an IGA score of 0 or 1 versus 45 (88.2% [76.1-95.6], p<0.0001) of 51 participants in the M1095 120mg augmented load treatment group. Odds ratio could not be calculated due to the placebo group containing no responders
Statistical Analysis 5: Comparison: Placebo vs Secukinumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; At Week 12, none (0.0% [95% CI 0.0-6.8]) of the 52 participants in the placebo group had an IGA score of 0 or 1 versus 41 (77.4% [63.8-87.7], p<0.0001) of 53 participants in the secukinumab 300mg treatment group. Odds ratio could not be calculated due to the placebo group containing no responders

2. Secondary Outcome: Number of Participants With a Psoriasis Area and Severity Index (PASI) Reduction of 100% (i.e. Clear of Psoriasis)
Description: PASI 100, i.e. a subject's psoriasis has completely cleared at Week 12, compared to baseline.
Time Frame: Week 12, as compared to Week 0 (baseline)
Measure: Count of Participants; unit: Participants
Groups:
- M1095 120mg - Regimen 1: M1095, 120 mg, given at Week 0, 2, 4, and 8 weeks.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- M1095 120mg - Regimen 2: M1095, 120 mg, given at Week 0, 2, 4, 6, 8, and 10 weeks.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- Placebo / M1095 120mg: Placebo, given at Week 0, 1, 2, 3, 4, 6, 8 and 10 weeks.
  Placebo: Placebo contains no active drug.
Arm/Group | M1095 30mg | M1095 60mg | M1095 120mg - Regimen 1 | M1095 120mg - Regimen 2 | Placebo / M1095 120mg | Secukinumab
Number analyzed (Participants) | 52 | 52 | 53 | 51 | 52 | 53
Participants | 9 | 13 | 20 | 17 | 0 | 15

3. Secondary Outcome: Number of Participants With a Psoriasis Area and Severity Index (PASI) Reduction of 90% (i.e. a 90% Improvement in Psoriasis)
Description: PASI 90, i.e. a subject's psoriasis has cleared by 90% at Week 12, compared to baseline
Time Frame: Week 12, as compared to baseline
Measure: Count of Participants; unit: Participants
Arm/Group | M1095 30mg | M1095 60mg | M1095 120mg - Regimen 1 | M1095 120mg - Regimen 2 | Placebo / M1095 120mg | Secukinumab
Number analyzed (Participants) | 52 | 52 | 53 | 51 | 52 | 53
Participants | 19 | 34 | 37 | 39 | 0 | 34

4. Secondary Outcome: Number of Participants With a Psoriasis Area and Severity Index (PASI) Reduction of 75% (i.e. a 75% Improvement in Psoriasis)
Description: PASI 75, i.e. a subject's psoriasis has cleared by 75% at Week 12, compared to baseline
Time Frame: Week 12, as compared to Week 0 (baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | M1095 30mg | M1095 60mg | M1095 120mg - Regimen 1 | M1095 120mg - Regimen 2 | Placebo / M1095 120mg | Secukinumab
Number analyzed (Participants) | 52 | 52 | 53 | 51 | 52 | 53
Participants | 34 | 46 | 45 | 46 | 0 | 48

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signing of the informed consent form i.e. the start of the screening period (Week -4) through to the end of the study (Week 52).
Description: Arms/groups for presentation of adverse event reporting were pre-specified in the Statistical Analysis Plan.
Groups:
- Placebo (Week 0 to Week 12): Placebo given at Weeks 0, 2, 4 and 8.
  Placebo: Placebo contains no active drug.
- M1095 30mg (Week 0 to Week 12): M1095, 30mg, given at Weeks 0, 2, 4 and 8.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- M1095 60 mg (Week 0 to Week 12): M1095, 60mg, given at Weeks 0, 2, 4 and 8.
  M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- M1095 120mg - Normal Load Group (Week 0 to Week 12): M1095, 120 mg, given at Weeks 0, 2, 4 and 8.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- M1095 120mg - Augmented Load Group (Week 0 to Week 12): M1095, 120 mg, given at Weeks 0, 2, 4, 6, 8 and 10.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- Secukinumab (Week 0 to Week 12): Secukinumab, 300mg, given at Weeks 0, 1, 2, 3, 4 and 8.
  Secukinumab: Secukinumab is a human immunoglobulin G1 (IgG1) monoclonal antibody that selectively binds IL-17A.
- M1095 - All Participants (Week 0 to Week 12 ): All participants receiving M1095, 30mg, 60mg, or 120mg from Week 0 to Week 12.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- M1095 - All Participants (Week 12 to Week 52): All participants receiving M1095, 30mg, 60mg, or 120mg from Week 12 to Week 44, including subjects randomised to placebo, who received M1095 120mg from Weeks 12, 14, 16, 20, etc.
  M1095: M1095 is a trivalent monomeric nanobody® that neutralizes interleukins IL-17A, IL-17F, and IL-17A/F.
- Secukinumab (Week 12 to Week 52): Secukinumab, 300mg, given at Weeks 12, 16, 20 and every 4 weeks to week 44)
  Secukinumab: Secukinumab is a human immunoglobulin G1 (IgG1) monoclonal antibody that selectively binds IL-17A.
Arm/Group | Placebo (Week 0 to Week 12) | M1095 30mg (Week 0 to Week 12) | M1095 60 mg (Week 0 to Week 12) | M1095 120mg - Normal Load Group (Week 0 to Week 12) | M1095 120mg - Augmented Load Group (Week 0 to Week 12) | Secukinumab (Week 0 to Week 12) | M1095 - All Participants (Week 0 to Week 12 ) | M1095 - All Participants (Week 12 to Week 52) | Secukinumab (Week 12 to Week 52)
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52 | 0/52 | 0/53 | 0/51 | 0/53 | 0/208 | 1/251 | 0/51
Serious Adverse Events (participants affected / at risk) | 1/52 | 2/52 | 1/52 | 1/53 | 1/51 | 0/53 | 5/208 | 12/251 | 2/51
Other Adverse Events (participants affected / at risk) | 11/52 | 13/52 | 16/52 | 18/53 | 15/51 | 14/53 | 62/208 | 57/251 | 16/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Week 0 to Week 12) (N=52) | M1095 30mg (Week 0 to Week 12) (N=52) | M1095 60 mg (Week 0 to Week 12) (N=52) | M1095 120mg - Normal Load Group (Week 0 to Week 12) (N=53) | M1095 120mg - Augmented Load Group (Week 0 to Week 12) (N=51) | Secukinumab (Week 0 to Week 12) (N=53) | M1095 - All Participants (Week 0 to Week 12 ) (N=208) | M1095 - All Participants (Week 12 to Week 52) (N=251) | Secukinumab (Week 12 to Week 52) (N=51)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroglycopenia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0 to Week 12) (N=52) | M1095 30mg (Week 0 to Week 12) (N=52) | M1095 60 mg (Week 0 to Week 12) (N=52) | M1095 120mg - Normal Load Group (Week 0 to Week 12) (N=53) | M1095 120mg - Augmented Load Group (Week 0 to Week 12) (N=51) | Secukinumab (Week 0 to Week 12) (N=53) | M1095 - All Participants (Week 0 to Week 12 ) (N=208) | M1095 - All Participants (Week 12 to Week 52) (N=251) | Secukinumab (Week 12 to Week 52) (N=51)
Nasopharyngitis (Infections and infestations) | 4 | 4 | 11 | 9 | 4 | 6 | 28 | 26 | 7
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 3 | 3 | 2 | 3 | 9 | 12 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 4 | 3 | 4 | 1 | 14 | 6 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 2 | 3 | 0 | 6 | 13 | 0
Headache (Nervous system disorders) | 1 | 0 | 3 | 3 | 1 | 3 | 7 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 1 | 2 | 0 | 6 | 5 | 2
Hypertension (Vascular disorders) | 2 | 3 | 1 | 0 | 2 | 1 | 6 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT03384745/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT03384745/SAP_001.pdf